CLINICAL TRIAL: NCT04340284
Title: Retrospective Study to Analyze Safety and Efficacy of Adipose Tissue Derived Stromal Vascular Fraction (SVF) Application in Treatment of Long Bones Nonunion
Brief Title: Adipose Tissue Derived Stromal Vascular Fraction (SVF) Application in Treatment of Long Bones Nonunion
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dr. Himanshu Bansal Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HimanshubansalFoundation
Record Dates: First submitted 2020-04-05; First posted 2020-04-09 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Nonunion of Fracture
MeSH Terms: conditions — Fractures, Ununited

STUDY DESIGN:
Intervention Model Description: retrospective study to report the outcome in patients treated with fluoroscopic guided per cutaneous injection of Adipose tissue derived stromal vascular fraction (SVF) at the site of fracture as an outpatient procedure between November 2012 to August 2018.
  The indication for this procedure was established atrophic non-union with no evidence of infection with maximum gap between the fragments to be<5 mm and duration not later than one year between the fracture and the procedure.
  Healing at the injury site was evaluated using clinical and radio logical examination at 1,2,6, and 12 months post-treatment.Anterior-posterior radio graphs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with nonunion of long bones (Experimental): A total of 11patients ( november 2012 to august 2018) with atrophic non-union of long bones already treated with percutaneous SVF implantation
  Interventions: Biological: autologous adipose tissue derived stromal vascular fraction (SVF)

INTERVENTIONS:
Biological: autologous adipose tissue derived stromal vascular fraction (SVF) — liquid and solid portion of lipo-aspirate after non enzymatic processing yields SVF.
  This isolation process yielded an abundant population of Adipose stromal cells(ASCs) which have multipotent differentiation potential. Immunophenotype is a CD14-, CD29+, CD31-, CD34low/+, CD45-, CD73+ and CD105+ ,
  , the SVF represents the 50-70% in volume of a lipoaspirate specimen. The SVF hosts a heterogeneous cell population (110x103 cells/ml on average) comprising mainly CD105+ mesenchymal stem cells (MSC, 20%), plus a wide number of CD34+ hematopoietic cells (40%).

SUMMARY:
Nonunion is a major complication of fractures.Per cutaneous bone marrow concentrate (BMC) application around fracture ends is being utilized with great success . Mesenchymal Stem Cells (MSCs)are one of the major cell types found in BMC responsible for results Adipose tissue is an alternative source for MSCs. Besides abundant and readily accessible it also overcomes issue of morbidity with bone marrow aspiration.

this retrospective analysis to report the outcome in patients treated with fluoroscopic guided percutaneous injection of SVF at the site of fracture as an outpatient procedure between November 2012 to August 2018.

DETAILED DESCRIPTION:
Nonunion is of major complication of fractures .The overall rate of non-union is still not clear but estimates from the published literature suggests a range between 5-10% of the total fractures.The gap in non-healing management has instigated the search for novel osteo-inductive substances. bone marrow concentrate is being utilized for many year with excellent results .Mesenchymal Stem Cells (MSCs)are one of the major cell types of the Bone Marrow Aspirate Concentrate (BMAC)that self-renovates and differentiates into multiple cell types of mesodermal origin such as osteoblasts, chondrocytes, and adipocytes.

Adipose tissue is an alternative source for MSCs .besides abundant and readily accessible it also overcomes issue of morbidity with bone marrow aspiration.

This retrospective analysis was conducted to report the outcome in patients treated with fluoroscopic guided percutaneous injection of SVF at the site of fracture as an outpatient procedure between November 2012 to August 2018.

The purpose of this study is to report the feasibility of minimally invasive percutaneous injection with autologous SVF and study the osteo-inductive efficacy of Adipose derived stromal cells in SVF in the management of non-union.

ELIGIBILITY:
Inclusion Criteria:

* Non-union or delayed union diagnosed after x-ray examination More than 4 cm distance from the joint

Exclusion Criteria:

* Multiple major fracture or untreated major fracture
* Infected fracture
* HIV, hepatitis B or hepatitis C infection at the time of screening
* Diagnosis of cancer
* Active treatment with immunosuppressive drugs or anticoagulant agents
* Known allergic reaction to components of study treatment and/or study injection

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Union | 8 weeks
  evidence of union on xray

SECONDARY OUTCOMES:
Short Form 12 survey | 1,2,6,12 months
  12 item questionnaire used to assess generic health outcomes. scores 0 to 100 with higher the better health

CONTACTS AND LOCATIONS:
Locations (1):
- Anupam Hospital, Rudrapur, Uttrakhand, India

IPD SHARING:
Plan to Share IPD: Yes
any information needed will be gladly shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: anytime
Access Criteria: email TO hbansal@drhbf.org
URL: http://www.drhbf.org

REFERENCES:
- [Result] Yoshimura K, Shigeura T, Matsumoto D, Sato T, Takaki Y, Aiba-Kojima E, Sato K, Inoue K, Nagase T, Koshima I, Gonda K. Characterization of freshly isolated and cultured cells derived from the fatty and fluid portions of liposuction aspirates. J Cell Physiol. 2006 Jul;208(1):64-76. doi: 10.1002/jcp.20636. PMID 16557516
- [Result] Caplan AI, Dennis JE. Mesenchymal stem cells as trophic mediators. J Cell Biochem. 2006 Aug 1;98(5):1076-84. doi: 10.1002/jcb.20886. PMID 16619257
- [Result] Prins HJ, Schulten EA, Ten Bruggenkate CM, Klein-Nulend J, Helder MN. Bone Regeneration Using the Freshly Isolated Autologous Stromal Vascular Fraction of Adipose Tissue in Combination With Calcium Phosphate Ceramics. Stem Cells Transl Med. 2016 Oct;5(10):1362-1374. doi: 10.5966/sctm.2015-0369. Epub 2016 Jul 7. PMID 27388241
- [Result] Saxer F, Scherberich A, Todorov A, Studer P, Miot S, Schreiner S, Guven S, Tchang LA, Haug M, Heberer M, Schaefer DJ, Rikli D, Martin I, Jakob M. Implantation of Stromal Vascular Fraction Progenitors at Bone Fracture Sites: From a Rat Model to a First-in-Man Study. Stem Cells. 2016 Dec;34(12):2956-2966. doi: 10.1002/stem.2478. Epub 2016 Sep 16. PMID 27538760